CLINICAL TRIAL: NCT01087749
Title: Pharmacokinetic Study of Propranolol, Losartan, and Eprosartan in Healthy Volunteers and Patients With Chronic Kidney Disease
Brief Title: Pharmacokinetic Study in Patients With Chronic Kidney Disease and Healthy Volunteers
Acronym: CKD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: PKUCSF2010
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Kidney Disease
MeSH Terms: conditions — Kidney Diseases | interventions — Propranolol; propranolol CR; Losartan; eprosartan; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronic Kidney Disease (Experimental): Propranolol, Losartan, and Eprosartan will be administered to patients who have been diagnosed with Chronic Kidney disease and have a glomerular filtration rate (GFR) below 40ml/min.
  Interventions: Drug: Propranolol; Drug: Losartan; Drug: Eprosartan
- Healthy Volunteers (Experimental): Propranolol, Losartan, and Eprosartan will be administered to healthy volunteers without chronic kidney disease.
  Interventions: Drug: Propranolol; Drug: Losartan; Drug: Eprosartan

INTERVENTIONS:
Drug: Propranolol — Propranolol 40mg PO will be given with 6oz of water.Blood samples will be obtained for 12 hours to determine the medication concentration in the plasma. There is no therapeutic effect on this study, since patients will receive a low single dose of the medication, and we'll assess the different pharmacokinetic parameters based on the concentrations of the medicine in plasma.
  Other Names: Propranolol Hydrochloride; Ciplar; Ciplar LA; Inderal; Inderal LA; Avlocardyl; Deralin; Dociton; Inderalici; InnoPran XL; Sumial; Anaprilinum; Bedranol SR
Drug: Losartan — Losartan 50mg PO will be given with 6oz of water. Blood samples will be obtained for 12 hours to determine the medication concentration in the plasma. There is no therapeutic effect on this study, since patients will receive a low single dose of the medication, and we'll assess the different pharmacokinetic parameters based on the concentrations of the medicine in plasma.
  Other Names: Cozaar; Losartan potassium; Anin
Drug: Eprosartan — Erythromycin 125mg PO will be given with 6oz of water. Blood samples will be obtained for 12 hours to determine the medication concentration in the plasma. There is no therapeutic effect on this study, since patients will receive a low single dose of the medication, and we'll assess the different pharmacokinetic parameters based on the concentrations of the medicine in plasma.
  Other Names: Teveten; Eprozar; Teveten HCT (paired with hydrochlorothiazide); Teveten Plus (paired with hydrochlorothiazide)

SUMMARY:
The purpose of this study is to find out how chemicals in the blood of patients with chronic kidney disease affect how medications are removed from the body. The patient will take one dose of three different drugs, one on each week, for a total of three single doses. The investigators want to find out if these three different medications are affected in different ways by the chemicals in the blood of patients with kidney disease.

DETAILED DESCRIPTION:
It has been demonstrated that proteins known as drug transporters in different human organs and tissues are important for a drug to be absorbed, distributed, metabolized, and eliminated (ADME)18. The chemical properties of drugs can affect whether it needs a transporter protein to enter the cell or not. It is not well known how these proteins are affected in chronic disease and how different drugs may be absorbed, metabolized, or eliminated differently in certain diseases. Preliminary studies suggest that some drugs (those requiring drug transporter proteins) may show altered elimination in the presence of uremic toxins. Uremic toxins are substances accumulated in the blood of patients with chronic kidney disease and many are not removed through hemodialysis (HD). We hypothesize that the different classes of drugs (BDDCS class1, 2, and 3) will have different degrees of changes in AUC, meaning that for a class 1 drug we would see less of a change in AUC than in a class 3 drug because a class 3 drug requires transporters. Previous studies can't make that comparison because they used different patients for each drug, so even if there were a change in a class 1 drug, it can't be compared to a class 3 drug. In order to get an accurate comparison, we will test the three drugs on the same patient and see how he AUC changes from drug to drug within the same patient comparing it to the healthy volunteer (taking the same three drugs).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18-70 years of age.
* Healthy volunteers or chronic kidney disease (GFR<40)
* Be able to provide written informed consent and comply with requirements of the study.
* Avoid eating grapefruit and drinking grapefruit juice from 7 days prior to the first study day until completion of the study.
* Abstinence from alcoholic beverages, caffeinated beverages and orange juice from 6pm the night before a study day until completion of the study day.
* Fast from food and beverages at least 8 hours prior to medication dosing.
* Be able to read, speak, and understand English.

Exclusion Criteria:

* Subjects with contraindications to taking the study drugs
* Subjects with known allergies to propranolol, losartan, or eprosartan.
* Subjects who smoke tobacco.
* Subjects with ongoing alcohol or illegal drug use.
* Subjects who are pregnant, lactating, or attempting to conceive.
* Subjects unable to maintain adequate birth control during the study.
* Subjects unable to follow protocol instructions or protocol criteria.
* Subjects with hematocrit < 30mg/dL.
* Subjects who are insulin requiring diabetics.
* Subjects with low, or low normal blood pressure (systolic blood pressure [BP] <100mmHg)
* Subjects with uncontrolled high blood pressure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | 3 weeks
  Three 12-hour days visits (on different weeks) will be investigated to obtain blood samples for 12 hours for three different medications. Blood samples will be obtained to determine the medication concentration in the plasma. There is no therapeutic effect on this study, since patients will receive a low single dose of the medication, and we'll assess the different pharmacokinetic parameters based on the concentrations of the medicine in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Z Benet, PhD, Principal Investigator — University of California, San Francisco; Lynda Frassetto, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Clinical Reserach Center, UCSF, San Francisco, California, United States

REFERENCES:
- [Background] Bianchetti G, Graziani G, Brancaccio D, Morganti A, Leonetti G, Manfrin M, Sega R, Gomeni R, Ponticelli C, Morselli PL. Pharmacokinetics and effects of propranolol in terminal uraemic patients and in patients undergoing regular dialysis treatment. Clin Pharmacokinet. 1976;1(5):373-84. doi: 10.2165/00003088-197601050-00004. PMID 1017154
- [Background] Lam JL, Shugarts SB, Okochi H, Benet LZ. Elucidating the effect of final-day dosing of rifampin in induction studies on hepatic drug disposition and metabolism. J Pharmacol Exp Ther. 2006 Nov;319(2):864-70. doi: 10.1124/jpet.106.108282. Epub 2006 Aug 11. PMID 16905688
- [Background] Lau YY, Okochi H, Huang Y, Benet LZ. Pharmacokinetics of atorvastatin and its hydroxy metabolites in rats and the effects of concomitant rifampicin single doses: relevance of first-pass effect from hepatic uptake transporters, and intestinal and hepatic metabolism. Drug Metab Dispos. 2006 Jul;34(7):1175-81. doi: 10.1124/dmd.105.009076. Epub 2006 Apr 19. PMID 16624870
- [Background] Lau YY, Huang Y, Frassetto L, Benet LZ. effect of OATP1B transporter inhibition on the pharmacokinetics of atorvastatin in healthy volunteers. Clin Pharmacol Ther. 2007 Feb;81(2):194-204. doi: 10.1038/sj.clpt.6100038. Epub 2006 Dec 27. PMID 17192770
- [Background] Guevin C, Michaud J, Naud J, Leblond FA, Pichette V. Down-regulation of hepatic cytochrome p450 in chronic renal failure: role of uremic mediators. Br J Pharmacol. 2002 Dec;137(7):1039-46. doi: 10.1038/sj.bjp.0704951. PMID 12429576
- [Background] Martin DE, Chapelsky MC, Ilson B, Tenero D, Boike SC, Zariffa N, Jorkasky DK. Pharmacokinetics and protein binding of eprosartan in healthy volunteers and in patients with varying degrees of renal impairment. J Clin Pharmacol. 1998 Feb;38(2):129-37. doi: 10.1002/j.1552-4604.1998.tb04401.x. PMID 9549643
- [Background] Michaud J, Naud J, Chouinard J, Desy F, Leblond FA, Desbiens K, Bonnardeaux A, Pichette V. Role of parathyroid hormone in the downregulation of liver cytochrome P450 in chronic renal failure. J Am Soc Nephrol. 2006 Nov;17(11):3041-8. doi: 10.1681/ASN.2006010035. Epub 2006 Oct 4. PMID 17021269
- [Background] Naud J, Michaud J, Leblond FA, Lefrancois S, Bonnardeaux A, Pichette V. Effects of chronic renal failure on liver drug transporters. Drug Metab Dispos. 2008 Jan;36(1):124-8. doi: 10.1124/dmd.107.018192. Epub 2007 Oct 16. PMID 17940133
- [Background] Nolin TD, Naud J, Leblond FA, Pichette V. Emerging evidence of the impact of kidney disease on drug metabolism and transport. Clin Pharmacol Ther. 2008 Jun;83(6):898-903. doi: 10.1038/clpt.2008.59. Epub 2008 Apr 2. PMID 18388866
- [Background] Sica DA, Halstenson CE, Gehr TW, Keane WF. Pharmacokinetics and blood pressure response of losartan in end-stage renal disease. Clin Pharmacokinet. 2000 Jun;38(6):519-26. doi: 10.2165/00003088-200038060-00005. PMID 10885588
- [Background] Sun H, Huang Y, Frassetto L, Benet LZ. Effects of uremic toxins on hepatic uptake and metabolism of erythromycin. Drug Metab Dispos. 2004 Nov;32(11):1239-46. doi: 10.1124/dmd.104.000521. Epub 2004 Jul 30. PMID 15286055
- [Background] Vanholder R, De Smet R, Glorieux G, Argiles A, Baurmeister U, Brunet P, Clark W, Cohen G, De Deyn PP, Deppisch R, Descamps-Latscha B, Henle T, Jorres A, Lemke HD, Massy ZA, Passlick-Deetjen J, Rodriguez M, Stegmayr B, Stenvinkel P, Tetta C, Wanner C, Zidek W; European Uremic Toxin Work Group (EUTox). Review on uremic toxins: classification, concentration, and interindividual variability. Kidney Int. 2003 May;63(5):1934-43. doi: 10.1046/j.1523-1755.2003.00924.x. PMID 12675874
- [Background] Wu CY, Benet LZ. Predicting drug disposition via application of BCS: transport/absorption/ elimination interplay and development of a biopharmaceutics drug disposition classification system. Pharm Res. 2005 Jan;22(1):11-23. doi: 10.1007/s11095-004-9004-4. PMID 15771225